CLINICAL TRIAL: NCT05701995
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Effect of Deucravacitinib on Quality of Life in Participants With Plaque Psoriasis in a Community Setting
Brief Title: A Study to Evaluate the Effect of Deucravacitinib on Quality of Life in Participants With Plaque Psoriasis in a Community Setting
Acronym: ARTISTYK
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IM011-237; U1111-1276-5158 (Registry Identifier: WHO)
Record Dates: First submitted 2023-01-16; First posted 2023-01-27 (Actual); Results first posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-08

CONDITIONS: Psoriasis
Keywords: plaque psoriasis; deucravacitinib; BMS-986165; Health related quality of life (HrQoL); QoL (quality of life); SOTYKTU
MeSH Terms: conditions — Psoriasis | interventions — deucravacitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Deucravacitinib (Experimental)
  Interventions: Drug: Deucravacitinib
- Placebo then Deucravacitinib (Placebo Comparator)
  Interventions: Drug: Deucravacitinib; Other: Placebo

INTERVENTIONS:
Drug: Deucravacitinib — Specified dose on specified days.
  Other Names: BMS-986165; Sotyktu
Other: Placebo — Specified dose on specified days.
  Arms: Placebo then Deucravacitinib

SUMMARY:
The purpose of this study is to evaluate the effect of deucravacitinib on quality of life (QoL) in participants with plaque psoriasis in a community setting.

ELIGIBILITY:
Inclusion Criteria

* Men and women diagnosed with stable plaque psoriasis for 6 months or more. Stable psoriasis is defined as no morphology changes or significant flares of disease activity in the opinion of the investigator.
* Deemed by the investigator to be a candidate for phototherapy or systemic therapy.
* ≥ 3% of Body Surface Area (BSA) involvement at the Screening Visit and Day 1
* Dermatology Life Quality Index (DLQI) score > 5 at the Screening Visit and Day 1
* Moderate-to-severe plaque psoriasis as defined by static Physician Global Assessment (s-PGA) ≥ 3 at the Screening Visit and Day 1

Exclusion Criteria:

Target Disease Exceptions:

* Non-plaque psoriasis (that is, guttate, pustular, erythrodermic, palmoplantar only involvement or drug-induced psoriasis) at Screening Visit or Day 1

Other protocol-defined inclusion/exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2023-01-31 (Actual); Primary Completion 2024-08-23 (Actual); Study Completion 2025-05-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (38):
- United States (35):
  - Local Institution - 0006, Phoenix, Arizona
  - Local Institution - 0034, Scottsdale, Arizona
  - Local Institution - 0015, North Little Rock, Arkansas
  - Local Institution - 0004, Bakersfield, California
  - Local Institution - 0009, Sacramento, California
  - Local Institution - 0022, San Diego, California
  - Local Institution - 0030, Centennial, Colorado
  - Local Institution - 0024, Washington D.C., District of Columbia
  - Local Institution - 0027, Brandon, Florida
  - Local Institution - 0016, Coral Gables, Florida
  - Riverchase Dermatology, Pembroke Pines, Florida
  - Local Institution - 0037, Atlanta, Georgia
  - Local Institution - 0020, Snellville, Georgia
  - Local Institution - 0007, Rolling Meadows, Illinois
  - Local Institution - 0025, Skokie, Illinois
  - Local Institution - 0036, Springfield, Illinois
  - Local Institution - 0003, Baton Rouge, Louisiana
  - Local Institution - 0018, Rockville, Maryland
  - Local Institution - 0010, Auburn Hills, Michigan
  - Local Institution - 0002, Waterford, Michigan
  - Local Institution - 0017, Las Vegas, Nevada
  - Local Institution - 0035, Reno, Nevada
  - Local Institution - 0032, New York, New York
  - Local Institution - 0013, New York, New York
  - Local Institution - 0001, Rochester, New York
  - Local Institution - 0005, Bexley, Ohio
  - Local Institution - 0012, Mayfield Heights, Ohio
  - Local Institution - 0019, Charleston, South Carolina
  - Local Institution - 0029, Cypress, Texas
  - Local Institution - 0028, Frisco, Texas
  - Local Institution - 0008, South Jordan, Utah
  - Local Institution - 0033, Springville, Utah
  - Local Institution - 0021, Bellevue, Washington
  - Local Institution - 0031, Mill Creek, Washington
  - Local Institution - 0014, Spokane, Washington
- Puerto Rico (3):
  - Local Institution - 0040, Caguas
  - Local Institution - 0038, Carolina
  - Local Institution - 0039, San Juan

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol-Myers Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 180 participants were randomized and of these 178 received at least one dose of study treatment.
Groups:
- BMS-986165 6mg QD: Participants received deucravacitinib at a dose of 6 mg daily (QD)
- Placebo: Participants received placebo daily (QD)
Period: Pre-Treatment
Arm/Group | BMS-986165 6mg QD | Placebo
Started (Started = Full Analysis Set/Randomized) | 120 | 60
Full Analysis Set Sub-population (All participants who were randomized to any treatment group with baseline static physician global assessment (s-PGA) >=3) | 107 | 49
Completed (Completed = Treated) | 119 | 59
Not Completed | 1 | 1
Not completed — Randomization Error | 1 | 1
Period: Treatment
Arm/Group | BMS-986165 6mg QD | Placebo
Started (Started = Treated) | 119 | 59
Completed | 104 | 49
Not Completed | 15 | 10
Not completed — Withdrawal by Subject | 8 | 4
Not completed — Lost to Follow-up | 2 | 3
Not completed — Adverse Event | 3 | 1
Not completed — Other Reason | 1 | 1
Not completed — Death | 1 | 0
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BMS-986165 6mg QD | Placebo | Total
Number analyzed (Participants) | 120 | 60 | 180
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.1 (14.92) | 47.5 (13.55) | 48.6 (14.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 20 | 68
  Male | 72 | 40 | 112
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 34 | 22 | 56
  Not Hispanic or Latino | 86 | 36 | 122
  Unknown or Not Reported | 0 | 2 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 1 | 6
  Black or African American | 3 | 6 | 9
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  White | 108 | 50 | 158
  Other | 2 | 3 | 5
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Dermatology Life Quality Index (DLQI) Score of 0 or 1 at Week 16
Description: Dermatology Life Quality Index (DLQI) is a participant-reported Quality of Life (QoL) survey which consists of 10 questions concerning symptoms and feelings, daily activities, leisure, work, school, personal relationships, and treatment during the last week. Each question is scored on a 4-point scale:
  0=not at all
  1. a little
  2. a lot
  3. very much The scores are added up to give a total score between 0 and 30. A lower total score means a better quality of life.
Time Frame: At Week 16
Population: Full Analysis Set: All Randomized Participants Full Analysis Set Sub-Population: All Randomized Participants with baseline static Physician Global Assessment ≥3 (s-PGA≥3)
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | BMS-986165 6mg QD | Placebo
Number analyzed (Participants) | 120 | 60
Percentage of Participants
  Full Analysis Set | 33.3 [25.0 to 42.5] | 6.7 [1.8 to 16.2]
  Full Analysis Set Sub-population: number analyzed (Participants) | 107 | 49
  Full Analysis Set Sub-population | 32.7 [24.0 to 42.5] | 6.1 [1.3 to 16.9]
Statistical Analysis 1: Comparison: BMS-986165 6mg QD vs Placebo; Full Analysis Set; Test type: Superiority; p = 0.0001, Stratified Cochran-Mantel-Haenszel (CMH); Odds Ratio (OR) = 7.7, 95% CI 2-sided [2.5 to 23.6]
Statistical Analysis 2: Comparison: BMS-986165 6mg QD vs Placebo; Full Analysis Set Sub-population; Test type: Superiority; p = 0.0003, Stratified Cochran-Mantel-Haenszel (CMH); Odds Ratio (OR) = 8.5, 95% CI 2-sided [2.4 to 30.4]

2. Secondary Outcome: Percentage of Participants Achieving a ≥ 4-point Reduction From Baseline in Dermatology Life Quality Index (DLQI) at Week 16
Description: The Dermatology Life Quality Index (DLQI) is a simple, 10-question survey used to measure the impact of skin conditions on a patient's quality of life. It assesses how much a skin condition affects various aspects of daily life, including symptoms, feelings, daily activities, work or school, personal relationships, and treatment.
  The DLQI is scored by summing the responses to its 10 questions. Each question is scored on a scale from 0 to 3:
  0 = Not at all
  1. = A little
  2. = A lot
  3. = Very much The total score ranges from 0 to 30, with higher scores indicating a greater impact on the patient's quality of life.
Time Frame: At Week 16
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | BMS-986165 6mg QD | Placebo
Number analyzed (Participants) | 120 | 60
Percentage of Participants
  Full Analysis Set | 72.5 [63.6 to 80.3] | 53.3 [40.0 to 66.3]
  Full Analysis Set Sub-population: number analyzed (Participants) | 107 | 49
  Full Analysis Set Sub-population | 72.9 [63.4 to 81.0] | 53.1 [38.3 to 67.5]
Statistical Analysis 1: Comparison: BMS-986165 6mg QD vs Placebo; Full Analysis Set; Test type: Superiority; p = 0.0107, Stratified Cochran-Mantel-Haenszel (CMH); Odds Ratio (OR) = 2.3, 95% CI 2-sided [1.2 to 4.4]
Statistical Analysis 2: Comparison: BMS-986165 6mg QD vs Placebo; Full Analysis Set Sub-population; Test type: Superiority; p = 0.0175, Stratified Cochran-Mantel-Haenszel (CMH); Odds Ratio (OR) = 2.3, 95% CI 2-sided [1.2 to 4.7]

3. Secondary Outcome: Change From Baseline in Whole-body Itch Numerical Rating Scale (NRS) Score at Week 16
Description: The whole-body itch Numerical Rating Scale (NRS) is a survey that participants fill out themselves. It uses an 11-point scale from 0 to 10, where 0 means 'no itch' and 10 means 'worst itch imaginable.' Participants indicate the severity of their itching from psoriasis by selecting the number that best describes the worst level of itching they experienced in the past 24 hours. A lower score means better outcomes, indicating less severe itching.
Time Frame: Baseline and at Week 16
Population: Full Analysis Set: Randomized Participants Full Analysis Set Sub-Population: Randomized Participants with baseline static Physician Global Assessment ≥3 (s-PGA≥3)
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | BMS-986165 6mg QD | Placebo
Number analyzed (Participants) | 120 | 59
Score on a Scale
  Full Analysis Set | -3.8 (2.86) | -1.8 (2.78)
  Full Analysis Set Sub-population: number analyzed (Participants) | 107 | 49
  Full Analysis Set Sub-population | -3.8 (2.73) | -1.8 (2.70)
Statistical Analysis 1: Comparison: BMS-986165 6mg QD vs Placebo; Full Analysis Set; Test type: Superiority; p < 0.0001, Covariance model; Adjusted Mean Difference = -2.0, 95% CI 2-sided [-2.9 to -1.2]
Statistical Analysis 2: Comparison: BMS-986165 6mg QD vs Placebo; Full Analysis Set Sub-population; Test type: Superiority; p < 0.0001, Covariance model; Adjusted Mean Difference = -2.2, 95% CI 2-sided [-3.0 to -1.3]

4. Secondary Outcome: Percentage of Participants With a Static Physician's Global Assessment (s-PGA) Score of 0 (Clear) or 1 (Almost Clear) With at Least a 2-point Reduction From Baseline at Week 16
Description: The Static Physician's Global Assessment (s-PGA) is a 5-point scale to evaluate the average severity of all psoriatic lesions based on redness, scaling, and thickness. The s-PGA measures psoriasis severity at a single point in time, without considering the initial condition. The scale rates the severity as clear (0), almost clear (1), mild (2), moderate (3), or severe (4). A lower score means better outcomes, indicating less severe psoriasis.
Time Frame: At Week 16
Population: All randomized participants with baseline static Physician Global Assessment ≥3 (s-PGA≥3)
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | BMS-986165 6mg QD | Placebo
Number analyzed (Participants) | 107 | 49
Percentage of Participants | 35.5 [26.5 to 45.4] | 8.2 [2.3 to 19.6]
Statistical Analysis 1: Comparison: BMS-986165 6mg QD vs Placebo; Full Analysis Set Sub-population; Test type: Superiority; p = 0.0004, Stratified Cochran-Mantel-Haenszel (CMH); Odds Ratio (OR) = 5.9, 95% CI 2-sided [2.0 to 17.4]

5. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) From Week 0 to Week 16
Description: An adverse event (AE) is defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in a clinical investigation participant administered study treatment that does not necessarily have a causal relationship with this treatment.
Time Frame: From Week 0 through Week 16
Population: As-treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-986165 6mg QD | Placebo
Number analyzed (Participants) | 119 | 59
Participants | 63 | 25

6. Secondary Outcome: Number of Participants With Treatment Emergent Serious Adverse Events (SAEs) From Week 0 to Week 16
Description: Serious Adverse Event (SAE) is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, and requires inpatient hospitalization or causes prolongation of existing hospitalization.
Time Frame: From Week 0 through Week 16
Population: As-treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-986165 6mg QD | Placebo
Number analyzed (Participants) | 119 | 59
Participants | 3 | 1

7. Secondary Outcome: Number of Participants With Laboratory Abnormalities in Potential Drug-Induced Liver Injury Tests From Week 0 to Week 16
Description: Number of participants with laboratory abnormalities in potential drug-induced liver injury tests.
  ALT=Alanine aminotransferase AST=Aspartate aminotransferase ULN=Upper limit of normal
Time Frame: From Week 0 through Week 16
Population: As-treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-986165 6mg QD | Placebo
Number analyzed (Participants) | 119 | 59
Participants
  ALT or AST > 3 X ULN | 1 | 0
  ALT or AST > 5 X ULN | 0 | 0
  Total Bilirubin > 2 X ULN | 0 | 0
  ALT or AST > 3 X ULN and Total Bilirubin > 2 X ULN on the same day | 0 | 0

8. Secondary Outcome: Number of Participants With Grade 3/ Grade 4 Laboratory Abnormalities From Week 0 to Week 16
Description: Blood samples were collected to assess the abnormalities in laboratory parameters. The laboratory parameters were graded by Common Terminology Criteria for Adverse Events (CTCAE). Grade 3=Severe; Grade 4=Life-threatening.
Time Frame: From Week 0 through Week 16
Population: As-treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-986165 6mg QD | Placebo
Number analyzed (Participants) | 119 | 59
Participants
  Hematology: Leukocytes (Grade 3) | 1 | 0
  Hematology: Platelets (Grade 4) | 1 | 0
  Chemistry: Potassium (Grade 3) | 1 | 0

9. Secondary Outcome: Number of Participants With Abnormalities in Vital Signs From Week 0 to Week 16
Description: Number of participants with abnormalities in vital signs including heart rate, systolic blood pressure, and diastolic blood pressure.
Time Frame: From Week 0 through Week 16
Population: As-treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-986165 6mg QD | Placebo
Number analyzed (Participants) | 118 | 58
Participants
  Heart Rate (Beats/Min): Value > 100 And Change From Baseline > 30 | 0 | 1
  Heart Rate (Beats/Min): Value < 55 And Change From Baseline < -15 | 0 | 0
  Heart Rate (Beats/Min): Not Reported | 0 | 0
  Systolic Blood Pressure (Mmhg): Value > 140 And Change From Baseline > 20 | 5 | 4
  Systolic Blood Pressure (Mmhg): Value < 90 And Change From Baseline < -20 | 0 | 0
  Systolic Blood Pressure (Mmhg): Not Reported | 0 | 0
  Diastolic Blood Pressure (Mmhg): Value > 90 And Change From Baseline > 10 | 19 | 6
  Diastolic Blood Pressure (Mmhg): Value < 55 And Change From Baseline < -10 | 0 | 1
  Diastolic Blood Pressure (Mmhg): Not Reported | 0 | 0

10. Secondary Outcome: Number of Participants With Clinically Significant Changes in Vital Signs From Week 0 to Week 16
Description: Vital Sign Measurements include: Body Temperature (C), Respiratory Rate (breaths/min), Seated Blood Pressure (mmHg) and Heart Rate (beats/min).
  Clinically significant changes in these measurements may need medical attention as they could indicate a potential health concern.
Time Frame: From Week 0 through Week 16
Population: As-treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-986165 6mg QD | Placebo
Number analyzed (Participants) | 119 | 59
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Participants were assessed for All-cause mortality, Serious adverse events and Other adverse events for up to approximately 20 months.
Description: All-cause mortality, serious adverse events (SAEs) and other adverse events were assessed in all-treated participants.
Arm/Group | BMS-986165 6mg QD | Placebo
All-Cause Mortality (participants affected / at risk) | 1/119 | 0/59
Serious Adverse Events (participants affected / at risk) | 3/119 | 1/59
Other Adverse Events (participants affected / at risk) | 32/119 | 12/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BMS-986165 6mg QD (N=119) | Placebo (N=59)
Angina pectoris (Cardiac disorders) | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 1 | 0
Death (General disorders) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BMS-986165 6mg QD (N=119) | Placebo (N=59)
COVID-19 (Infections and infestations) | 7 | 2
Nasopharyngitis (Infections and infestations) | 8 | 2
Sinusitis (Infections and infestations) | 6 | 0
Upper respiratory tract infection (Infections and infestations) | 4 | 3
Headache (Nervous system disorders) | 2 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Acne (Skin and subcutaneous tissue disorders) | 9 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-25): https://cdn.clinicaltrials.gov/large-docs/95/NCT05701995/Prot_SAP_000.pdf